CLINICAL TRIAL: NCT04840576
Title: Prophylactic Negative Wound Pressure Therapy (PICO-7) Following Surgery for Revascularization of Patients With Chronic Lower Limb Ischemia (PICO-Vasc Study): A Prospective Ramdomised Clinical Trial
Brief Title: Prophylactic Negative Wound Pressure Therapy (PICO-7) Following Groin Incisions in Vascular Surgery (PICO-Vasc Study)
Acronym: PICO-Vasc
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Kerbi Alejandro Guevara-Noriega, Sabadell, Parc Tauli, Spain (Unknown); Elena Gonzalez Canas, Sabadell, Parc Tauli, Spain (Unknown); Marta Camats Terre, Sabadell, Parc Tauli, Spain (Unknown); Eduardo Arrea Salto, Sabadell, Parc Tauli, Spain (Unknown); Antonio Giménez Gaibar, Sabadell, Parc Tauli, Spain (Unknown); Marta Santos Espi, Sabadell, Parc Tauli, Spain (Unknown)
Responsible Party: Principal Investigator, Laura Rodriguez-Lorenzo, Vascular and Endovascular Surgeon, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TauliCV002
Record Dates: First submitted 2021-03-24; First posted 2021-04-12 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Surgical Wound Infection
Keywords: Surgical Wound Infection; Seroma; Hematoma; Lymphorrhagia; Lymphocele; Extended Hospital Admission; Postoperative Mortality
MeSH Terms: conditions — Surgical Wound Infection; Seroma; Hematoma; Lymphocele

STUDY DESIGN:
Intervention Model Description: 2 parallel groups receiving different interventions
Who Masked: Participant
Masking Description: Once it is confirmed that the patient meets the inclusion criteria, exclusion criteria have been ruled out and after signing the corresponding informed consent, randomization will be carried out. The randomization will be carried out by the research center, and the assignment will be made through opaque envelopes.
  The assignment of the intervention group will be made by the nursing staff of the surgical area.
  In cases where a bilateral inguinal approach coexists in the same surgical procedure, the right side will be randomized; the contralateral incision will receive alternative therapy by default.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Dressing (Placebo Comparator): waterproof sterile dressing OPSITE Post-Op Visible, Smith & Nephew, UK
  Interventions: Other: Regular waterproof sterile dressing.
- Prophylactic negative wound pressure dressing (Experimental): PICO-7, Smith & Nephew, UK
  Interventions: Other: Prophylactic Negative Pressure Dressing

INTERVENTIONS:
Other: Regular waterproof sterile dressing. — Waterproof sterile dressing OPSITE Post-Op Visible, Smith & Nephew, UK
  Arms: Conventional Dressing
Other: Prophylactic Negative Pressure Dressing — Negative wound pressure dressing: PICO-7, Smith & Nephew, UK
  Arms: Prophylactic negative wound pressure dressing

SUMMARY:
Comparison between waterproof sterile dressing OPSITE Post-Op Visible, Smith & Nephew, UK and PICO-7, Smith & Nephew, UK in terms of inguinal surgical wound infection and complications after lower limb revascularization.

DETAILED DESCRIPTION:
Patients will follow a preoperative preparation:

* Routine pre-surgical skin hygiene with soap or antiseptic agent
* Groin shaving with a machine
* Preoperative antibiotic prophylaxis with cefazolin 2 gr ev. single dose or clindamycin 900 mg ev. in case of allergy to beta-lactams 30 min before the start of the intervention. In case of prolongation of the intervention (> 4h), a second antibiotic dose will be administered
* Surgical field antisepsis using a sterile swab soaked in 2% chlorhexidine solution in 70% isopropyl alcohol, except for contraindications (such as potential contact with mucosa or open wounds, in which case 10% povidone-iodine solution will be used); usual sizing.

At the end of the revascularization surgical procedure, the inguinal wound will be closed using 2-0 or 3-0 Vicryl subcutaneous absorbable suture (Ethicon Inc, Somerville, NJ, USA) in two independent planes and skin closure with metal staples (B / Braun Manipler® AZ). The opaque randomization result allocation envelope will then be opened and the surgical area nurse will cover the wound with one of the two assigned dressings:

* Group 1 (intervention group): The surgical wound will be covered in a sterile manner with prophylactic TPN (PICO-7, Smith & Nephew, UK).
* Group 2 (control group): The surgical wound will be covered in a sterile way with the usual dressing (waterproof sterile dressing OPSITE Post-Op Visible, Smith & Nephew, UK).

During admission, regular follow-up will be carried out. On the 7th day, the dressings of both groups will be lifted. From this moment, if the wound allows it, air healing will be carried out without new dressings. After discharge from the hospital, the surgical wound evaluation will be carried out by the nurse responsible for Outpatient Consultations at 14 and 30 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-90
* Undergoing elective revascularization surgery (Rutherford clinical categories 4-6 / Fontaine III and IV) requiring a longitudinal inguinal approach (a longitudinal inguinal incision is defined as the one that runs from the inguinal ligament to the femoral bifurcation, performed with the intention of approaching the vascular bundle).
* Surgery performed by investigator and co-investigators: Vascular Surgeons of the Vascular Surgery Department at the Parc Taulí Hospital.
* Patients must be able to understand the study and sign the specific informed consent before surgery.

Exclusion Criteria:

* Urgent surgery
* Interventions in which transverse groin wounds.
* Presence of active groin infection that prevents primary closure
* Pediatric patients, pregnant women or patients with impaired higher functions who cannot understand the study or collaborate with its protocolized follow-up.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Surgical Wound Infection Rate | 30 days
  Number of participant with surgical wound with inflammatory signs according to the treating surgeon criteria in the first 30 days.

SECONDARY OUTCOMES:
Surgical Wound Complications Rate | 30 days
  Number of participant with surgical wound complications according to medical criteria of any of the following signs:
  * Seroma or lymphocele
  * Surgical wound dehiscence
  * Hematoma
  * Lymphorrhagia To be measured in 30 days.
Seroma or lymphocele rate | 30 days
  Number of participant with subcutaneous non-hematic liquid collection in the surgical bed of a closed wound. Its suspicion according to medical criteria will require puncture drainage and microbiological culture in 30 days after surgery
Surgical wound dehiscence rate | 30 days
  Number of participant with separation of the edges of part or all of a previously sutured wound in the 30 days after surgery
Rate of Hematoma | 30 days
  Number of participant with blood collection organized in the surgical bed of a closed wound in the 30 days after surgery
Rate of Lymphorrhagia | 30 days
  Number of participant with discharge of clear fluid through a surgical wound in the 30 days after surgery
Extended hospital admission rate | 30 days
  Number of participant with prolonged admission of more than 14 days due to cause/s related to the inguinal surgical wound complications or the need for reoperation, as well as, hospital readmission due to problems related to the inguinal surgical wound
Postoperative mortality Rate | 30 days
  Rate of death in the 30 days after surgery
Surgical wound infection-related mortality Rate | 30 days
  Rate of mortality secondary to infection of the surgical wound or due to causes related to complications of the inguinal surgical wound.
Level of postoperative pain | 7 days
  Measurement of postoperative pain in the 7 days after surgery. Carried out using the visual analog scale (VAS) applied to the patient

CONTACTS AND LOCATIONS:
Overall Officials: Kerbi A Guevara Noriega, MD MSc PhD, Study Chair — Vascular and Endovascular Surgery
Locations (1):
- Consorcio Sanitario Parc Tauli - Hospital Universitario., Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Correia RM, Nakano LC, Vasconcelos V, Cristino MA, Flumignan RL. Prevention of infection in peripheral arterial reconstruction of the lower limb. Cochrane Database Syst Rev. 2025 Oct 29;10(10):CD015022. doi: 10.1002/14651858.CD015022.pub2. PMID 41159585
- [Derived] Rodriguez Lorenzo L, Salto EA, Gonzalez Canas E, Madrazo Gonzalez Z, Espi MS, Gimenez Gaibar A. Incisional Negative Pressure Wound Therapy After Revascularisation Surgery in Patients with Peripheral Arterial Disease: A Randomised Trial (PICO-Vasc Study). Eur J Vasc Endovasc Surg. 2024 Aug;68(2):238-244. doi: 10.1016/j.ejvs.2024.04.031. Epub 2024 Apr 25. PMID 38677468